CLINICAL TRIAL: NCT06671041
Title: Treating Lid Wiper Epitheliopathy With Perfluorohexyloctane
Brief Title: Treating Lid Wiper Epitheliopathy
Acronym: TLWE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-03-01AS
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye; Visual Acuity
Keywords: Optometry; Dry Eye; Lens Wiper
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Preservative-free eye drop (Experimental): Participants were assigned to use a preservative-free eye drop 4X a day
  Interventions: Drug: Preservative Free eye drop

INTERVENTIONS:
Drug: Preservative Free eye drop — Participants were required to use a lubricating eye drop

SUMMARY:
Lid wiper epitheliopathy (LWE) is a relatively new entry into the abundance of clinical ocular surface health signs. LWE was first reported in 2002 as a potential cause for dry eye disease (DED) (Korb et al., 2002). This clinical sign is visualised by everting the eyelid after a dye has been applied and observing the palpebral conjunctiva proximal to the eyelashes

DETAILED DESCRIPTION:
Lid wiper epitheliopathy (LWE) is a relatively new entry into the abundance of clinical ocular surface health signs. LWE was first reported in 2002 as a potential cause for dry eye disease. This clinical sign is visualised by everting the eyelid after a dye has been applied and observing the palpebral conjunctiva proximal to the eyelashes. An observable line at the mucocutaneous junction, called the line of Marx, is present in all eyelids and any further staining of the tissue in the palpebral marginal conjunctiva can be regarded as LWE. LWE has been described as a micro-trauma caused by inadequate ocular lubrication and/or excessive friction. The lid wiper is one of the most sensitive conjunctival tissue areas of the ocular surface and upper eyelid LWE has been reported to be highly correlated to ocular surface discomfort and DED

Korb, theorised some plausible aetiologies for LWE. They were all ultimately linked to frictional related damaged initiated by 1) tear film dysfunction not including tear volume (since normal Schirmer testing was an inclusion in their study), 2) localised disorders of the lid wiper itself, 3) aberrant blinking, 4) ocular surface abnormalities at the cellular level (subclinical) to initiate excessive localised trauma, and 5) conditions that would lead to inflammation of the lid wiper.

The TFOS executive summary determined that a complete review of the clinical trials revealed a potential link of LWE to DED and suggested that future trials be performed to make conclusions as to which interventions might deliver the greatest impact Because LWE has been linked to DED, most of the proposed treatment strategies to relieve LWE have paralleled after treatments for DED and MGD. Treatment options fall into several categories. They are as follows: blinking, tear supplements and lubricants, tear retention agents, tear stimulants (secretagogues), biological tear substitutes, anti-inflammatory therapy, essential fatty acids, treatment of MGD and environmental strategies (including in-office treatments).

Excessive tear evaporation due to a deficient lipid layer is believed to be the most common cause of DED, and most evaporative DED is associated with MGD. Perfluorohexyloctane (PFHO) ophthalmic solution (MIEBO™; Bausch + Lomb) is a preservative-free eye drop that has demonstrated the ability to form a long-lasting barrier that inhibits evaporation in preclinical studies. FDA approval of PFHO was based on results from 2 pivotal clinical trials (GOBI [NCT04139798] and MOJAVE [NCT04567329]) in patients with DED and clinical signs of MGD, which demonstrated consistent improvements in both signs and symptoms of DED (Karpecki et al., 2023; Vittitow et al., 2023). PFHO is the first and only FDA-approved eye drop that directly targets tear

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* best corrected visual acuity (BCVA) of 20/100 or better
* who have symptomatic DED will be recruited (SPEED ≥6)
* Subjects will also be required to have a LWE score of 1.0 or greater to be included in the study.
* Subjects will be required to discontinue contact lens wear throughout the study.

Exclusion Criteria:

* known systemic health conditions that are known to alter tear film physiology (e.g., primary and secondary Sjögren's syndrome),
* have a history of ocular surgery within the past 12 months, have a history of severe ocular trauma, active ocular infection or inflammation,
* are currently using Accutane or ocular medications, or if they are pregnant or breast feeding.
* Artificial tear use will be discontinued at least one week prior to enrollment. Subjects with a condition or in a situation, which in the examiner's opinion, may put the subject at significant risk, may confound the study results, or may significantly interfere with their participation in the study will be excluded.
* Subjects that have had a physical meibomian gland treatment withing 1 month of enrollment (iLux, Lipiflow, etc.) will be excluded.
* Subjects will not be allowed to use any eye drops beyond their assignment during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
VAS | 2-Months
  VAS on a scale from 0-100 will be reported at baseline, 2 weeks, 1 month and 2 months and recoreded to see if there is a reduction in the percentage of subjects with a reduction in VAS scores for eye dryness, eye scratchiness, eye gritty/sandy feeling, eye irritation/soreness, eye burning/stinging, tired eyes, and itchy eyes (0-100)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Maitland Vision Center, Orlando, Florida
  - Complete Eye Care of Medina, Medina, Minnesota
  - Montaquila, Warwick, Rhode Island
  - The Southern College of Optometry, Memphis, Tennessee

REFERENCES:
- [Derived] Lievens C, Pucker AD, Franklin Q, Montaquila SM, Giedd B, Wesley G, Bromley M, Coker Z, Meyers J, Vianya-Estopa M. Investigating the Effect of Reducing the Signs and Symptoms of Lid Wiper Epitheliopathy in Patients With Dry Eye Disease With Perfluorohexyloctane. Curr Ther Res Clin Exp. 2025 Mar 20;102:100786. doi: 10.1016/j.curtheres.2025.100786. eCollection 2025. PMID 40276144